CLINICAL TRIAL: NCT00161772
Title: Double-blind, Randomized, Multicenter Dose-finding Study to Investigate the Safety and Immunogenicity of Two Vaccinations With FSME IMMUN NEW in Healthy Volunteers Aged 1 to 6 Years.
Brief Title: Dose-finding Study to Investigate the Safety and Immunogenicity of Two Vaccinations With FSME IMMUN NEW in Healthy Volunteers Aged 1 to 6 Years.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 199
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Tick-borne Encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne

INTERVENTIONS:
Biological: Tick-borne Encephalitis Vaccine

SUMMARY:
The purpose of this study is to investigate the safety and immunogenicity of three different concentrations of a TBE vaccine in healthy children aged 1 to 6 years.

ELIGIBILITY:
Inclusion Criteria:

Male and female children will be eligible for participation in this study if:

* they are 1 year (from the 1st birthday) to 6 years (to the last day before the 6th birthday) old;
* they are clinically healthy;
* their legal representative understands the nature of the study, agrees to its provisions and gives written informed consent;
* their legal representative agrees to keep a Volunteer Diary.

Exclusion Criteria:

Children will be excluded from participation in this study if they:

* have a history of any previous TBE vaccination;
* have a history of TBE infection or show evidence of a latent TBE infection (as demonstrated by screening ELISA > 126 VIEU/ml and / or neutralization test > 1:10);
* have a history of allergic reactions, in particular to one of the components of the vaccine;
* have received antipyretics within 4 hours prior to the first TBE vaccination;
* suffer from a disease that cannot be effectively treated or stabilized;
* suffer from a disease (e.g. autoimmune disease) or are undergoing a form of treatment that can be expected to influence immunological functions;
* suffer from chronic, degenerative and / or inflammatory disease of the central nervous system;
* are known to be HIV positive (a special HIV test is not required for the purpose of the study);
* suffer from a febrile illness at study entry;
* have a history of vaccination against yellow fever and / or Japanese B-encephalitis;
* are participating simultaneously in another clinical trial.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2002-03; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Behre, MD, Principal Investigator — Hauptstrasse 240, 77694 Kehl, Germany
Locations (23):
- Grieskirchner Strasse 17, Wels, Austria
- Germany (22):
  - Neuschwansteinstrasse 5, Augsburg
  - Marktplatz 3, Bad Saulgau
  - Hauptstrasse 9, Bietigheim-Bissingen
  - Salzgasse 11, Calw
  - Mohrenstrasse 8, Coburg
  - Bahnhofstrasse 1, Elzach
  - Rheinstrasse 13, Ettenheim
  - Peter-Seifert-Strasse 5, Gersfeld
  - Solothurner Strasse 2, Heilbronn
  - Hauptstraße 240, Kehl
  - Schwarzwaldstrasse 20, Kirchzarten
  - Altoettingerstrasse 3, Landsberg
  - Rastatter Strasse 7, Mannheim-Secken
  - Heubischer Strasse 39, Neustadt/Cbg
  - Dohmbuehlerstrasse 8, Nuremberg
  - Glogauer Strasse 15, Nuremberg
  - Tuchbergstrasse 2, Oberndorf / Neckar
  - Wilhelmstrasse 7, Offenburg
  - Asternweg 11a, Offenburg
  - Berneckstrasse 19, Schrammberg
  - Hauptstrasse 11, Tegernsee
  - Broner Platz 6, Weingarten